CLINICAL TRIAL: NCT06616545
Title: French Observatory for Patients with Type 3 Glycogenosis
Status: Recruiting | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Other Study IDs: GSD3 French Registry
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Glycogen Storage Disease Type III
MeSH Terms: conditions — Glycogen Storage Disease Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glycogen Storage Disease Type III

SUMMARY:
Glycogen storage disease type III (GSD-III) or Cori/Forbes disease, is caused by autosomal recessive mutations in the AGL gene, which codes for the glycogen debranching enzyme (GDE) involved in the release of glucose-1P from glycogen branches. Abnormal glycogen accumulation is responsible for frequent hypoglycaemia and symptoms in the liver and striated muscles (GSD-IIIa), although some patients present with liver involvement only (GSD-IIIb). In childhood, the phenotype is mainly characterised by hepatomegaly, short stature and hypoglycaemia, with minimal skeletal muscle involvement. While liver symptoms improve spontaneously around puberty, skeletal muscle weakness develops progressively in adulthood and becomes a major feature of GSD-IIIa.

Currently, there is no treatment other than dietary management tailored to the individual to limit glycogen storage and avoid hypoglycaemia.

The French GSD-III registry is a multicentre online registry dedicated to patients with type III glycogen storage disease followed in France. It has been approved by ethical and regulatory authorities. Its main inclusion criteria is the presence of a proven pathogenic AGL gene mutation and/or reduced glycogen debranching enzyme activity.

The aims of the registry are to provide a tool for recording detailed diagnostic, metabolic, neurological, cardiac and biological data on French patients with GSD-III, so as to enable i) a precise natural history of the disease, ii) identification of the outcome measures most sensitive to disease progression, iii) assessment of the frequency of the various complications of the disease and iv) identification of prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with molecularly characterised Glycogen Storage Disease Type III

Exclusion Criteria:

* Patients diagnosed with GSD type 3 refusing to take part in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GSD type 3 patients from French national reference centres
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fasting period | Through study completion, an average of 10 years
  Measuring changes in the duration of the fasting period

SECONDARY OUTCOMES:
6MWT distance | Through study completion, an average of 10 years
  Measurement of changes in distance covered in the 6-minute walk test.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Aphp Antoine Beclere, Clamart
  - CHU du Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Institue of Myology, Paris